CLINICAL TRIAL: NCT04776343
Title: Prospective, Randomized Study Comparing Two Populations of Patients Treated With Anti VEGF for Diabetic Macular Edema, One Being Followed at the Hospital and the Other One Being Followed at Home Using a Software Allowing Self-assessment of Visual Acuity
Brief Title: Study Comparing Two Populations of Patients Treated With Anti VEGF for Diabetic Macular Edema, One Being Followed at the Hospital and the Other One Being Followed at Home Using a Software Allowing Self-assessment of Visual Acuity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020_06_02
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedecine follow-up (Experimental)
  Interventions: Other: telemedecine follow-up
- Hospital follow-up (No Intervention)

INTERVENTIONS:
Other: telemedecine follow-up — weekly home-based follow-up of visual acuity on electronic tablet
  Arms: Telemedecine follow-up

SUMMARY:
Verify the reliability of VA measured every week at home, by the patient using a TC, compared to the reliability of VA also measured by the patient using a TC but every 2 month at the hospital, during standard DME follow-up visits

ELIGIBILITY:
Inclusion Criteria:

Will be included in the study, patients with all of the following criteria:

* aged ≥ 25 years old (the minimum age is set at 25 years old in order to include patient with controlled diabetes);
* diagnosed with DME;
* followed and treated by anti-VEGF IVT in the ophthalmology debarment at Hopital Saint Joseph Marseille;
* having a VA score ≥ 20/100;
* able to understand the study and to use a TC;
* having an internet access at home;
* having given free and informed written consent;
* being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

Will not be included in the study, patients with one of the following criteria:

* treated for another pathology that DME;
* already participating to another research study;
* pregnant or breastfeeding woman;
* subject to a measure for the protection of justice.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with VA evolution in the two groups | 36 months
  rate in percentage

SECONDARY OUTCOMES:
Variation of the VA measured using ETDRS scale on TC for the patients followed at home | 36 months
Variation of the VA measured using ETDRS scale on TC for the patients followed at the hospital | 36 months
Number of follow-up and injection visits for each patient according to their group | 36 months
Average time between the follow-up visit and the IVT (if performed) | 36 months
  in days
Variations in foveolar thickness and maximum central retinal thickness on OCT | 36 months
Change in quality of life for patients in group 1 compared to group 2 | 36 months
  the quality of life is assessed with EQ-5D-5L questionnaire
Change in the total cost per patient for patient in group 1 compared to group 2. | 36 months
  The total cost per patient is calculated from the number of follow-up visits, the number of procedures (OCT and fundus retinography) and the number of IVTs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Joseph Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No